CLINICAL TRIAL: NCT04998994
Title: The Effects of Wheat Sprouts Supplements on the Key Health Indicators of the Patients With Breast Cancer After Chemotherapy
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Quzhou Kecheng People's Hospital (Unknown); Beijing Shijitan Hospital, Capital Medical University (Other); Jinhua Municipal Central Hospital (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-172
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2019-05

CONDITIONS: Nutritional Status, Immune Function, Quality of Life Uring the Progress of Chemotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: wheat sprouts supplement — Maiji tablets, a wheat sprouts supplement, were used to treat 26 patients during the progress of chemotherapy

SUMMARY:
To explore the effects of wheat sprouts supplements on the key health indicators of the patients with breast cancer after chemotherapy, Maiji tablets, a wheat sprouts supplement, were used to treat 26 patients during the progress of chemotherapy and nutritional status, immune function, quality of life were measured and evaluated. Through data analysis, we found that Maiji tablets may improve the symptoms of appetite loss, nausea and vomiting, and fatigue in patients with breast cancer during chemotherapy. Meanwhile it may help patients maintain weight, keep appetite and improve the food intake.

ELIGIBILITY:
Inclusion Criteria:

- patients diagnosed with breast cancer, receiving chemotherapy for the first time

Exclusion Criteria:

- Patients with severe liver or kidney disease or other infectious diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with breast cancer, receiving chemotherapy for the first time
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
quality of life | 28 days
  Quality of life was measured by quality of life assessment form
weight | 28 days
  the weight of patients
nutritional status | 28 days
  nutritional status of patients

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No